CLINICAL TRIAL: NCT05379621
Title: Socio-economic, Meteorological and Environmental Factors Associated With the Incidence of COVID-19 in the Alpes-Maritimes and the City of Nice
Brief Title: Socio-economic, Meteorological and Environmental Factors Associated With the Incidence of COVID-19
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22DSP01
Record Dates: First submitted 2022-05-16; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: COVID-19 infection — All persons of legal age or not resident in the Alpes-Maritimes between 03/01/2021 and 14/02/2021 with a COVID-19 diagnosis.

SUMMARY:
Socio-demographic factors in relation to the diagnosis of COVID cases are increasingly mentioned in the role of transmission, but unfortunately with a small number of conclusive publications on French data. Our objective is to analyse the distribution of cases according to these factors and their possible role during the first 6 weeks of 2021 when the Alpes Maritimes was the department with the highest incidence rate. The collaboration between ARS06 and the Public Health Department in the field of COVID-19 has made it possible to have a departmental bulletin for monitoring the evolution of the epidemic (incidence, screening, hospitalisation). Knowledge of the socio-demographic, meteorological and environmental factors associated with the transmission of SARS-CoV2 would make it possible to reflect on how to act on these factors and to implement a public health policy.

ELIGIBILITY:
Inclusion Criteria:

Any person, adult or not, residing in the Alpes-Maritimes between 03/01/2021 and 14/02/2021 with a COVID-19 diagnosis.

Exclusion Criteria:

Non resident in the Alpes-Maritimes

Ages: 0 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population of legal age or not residing in the Alpes Maritimes department between 03/01/2021 and 14/02/2021, i.e. 1078729 inhabitants in the Alpes Maritimes, including 342979 in the city of Nice
Sampling Method: Non-Probability Sample
Enrollment: 28377 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2021-02-14 (Actual); Study Completion 2021-02-14 (Actual)

PRIMARY OUTCOMES:
Weekly incidence rate of COVID-19 in the Alpes-Maritimes during the study period. | Between 03/01/2021 and 14/02/2021
  Weekly incidence rate in the Alpes Maritimes according to the age group, by district of Nice and town

SECONDARY OUTCOMES:
Weekly incidence rate of COVID-19 in the Alpes-Maritimes during the study period according to participants' social and economic factors | Between 03/01/2021 and 14/02/2021
  Weekly incidence rate by social disadvantage index and others socioeconomic indicators by Census block of Nice, correlation analyses
Weekly incidence rate of COVID-19 in the Alpes-Maritimes during the study period according to climatic factors | Between 03/01/2021 and 14/02/2021
  Correlation of incidence rates with temperature, humidity, concentrations in air pollutants (fine particles, nitrogen oxides)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, France

REFERENCES:
- [Derived] Marine Barjoan E, Chaarana A, Festraets J, Geloen C, Prouvost-Keller B, Legueult K, Pradier C. Impact of social and demographic factors on the spread of the SARS-CoV-2 epidemic in the town of Nice. BMC Public Health. 2023 Jun 6;23(1):1098. doi: 10.1186/s12889-023-15917-z. PMID 37280635